CLINICAL TRIAL: NCT05231473
Title: Impact Of The Nurse Enhanced Recovery After Surgery Coordinator On The Compliance Of Multimodal Rehabilitation Programs In Colorectal Surgery (nursERAS-BCN)
Brief Title: Impact Of The Nurse Enhanced Recovery After Surgery Coordinator On The Compliance In Colorectal Surgery (nursERAS-BCN)
Acronym: nursERAS-BCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, José Antonio Jerez González, Enhanced Recovery After Surgery Coordinator, Hospital Universitari de Bellvitge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR426/21
Record Dates: First submitted 2022-01-11; First posted 2022-02-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: ERAS; Enhanced Recovery; Compliance, Treatment; Compliance, Patient; Nurse's Role; Colon Disease; Rectum Disease
MeSH Terms: conditions — Patient Compliance; Colonic Diseases; Rectal Diseases

STUDY DESIGN:
Intervention Model Description: This study is designed as a quasi-experimental study with a control group, an intervention group, without random assignment and multicenter trial; which is carried out at two centers in Barcelona, Spain: Bellvitge University Hospital (BUH) and Hospital Germans Trias i Pujol (HGTiP), between December 2021 and November 2023. The participants are assigned according to the implanted and functioning program of each center, to one of two arms: a control arm, in which they join the ERAS program without NEC (group I), and an intervention arm, in which the participants will be included in the ERAS program with NEC (group II).
  In HGTiP, the ERAS program without NEC is carried out in a standardized way, and in BUH it is carried out with NEC for all patients. The study directly compares both programs and their compliance in patients who are candidates for elective colorectal surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (No Intervention): The participants are assigned according to the implanted and functioning program of each center. In this case, without Nurse Enhanced Recovery After Surgery Coordinator. It will be the control group. ERAS program will be working without this role.
- Nurse Coordinator (Experimental): The participants are assigned according to the implanted and functioning program of each center. In this case, with Nurse Enhanced Recovery After Surgery Coordinator. It will be the intervention group. ERAS program will be working with this role.
  Interventions: Other: Nurse Enhanced Recovery After Surgery participation

INTERVENTIONS:
Other: Nurse Enhanced Recovery After Surgery participation — Bellvitge University Hospital will include the NEC participation along Enhanced Recovery After Surgery program.
  Other Names: NEC participation
  Arms: Nurse Coordinator

SUMMARY:
Purpose. The aim of this study is to evaluate the impact of the implementation of the Nurse Enhanced Recovery After Surgery Coordinator (NEC), within the Enhanced Recovery After Surgery (ERAS) program, in relation to the compliance of patients undergoing colorectal surgery.

Methods. Quasi-experimental study with a control group, an intervention group and without random assignment in a multicenter trial; between December 2021 and November 2023. Patients older than 18 years with planned elective intervention of major colorectal surgery will be included; excluding those without social support, with psychiatric illness, cognitive difficulty, planning of simultaneous or emergency surgery. In the intervention arm they will have NEC and in the control group they will not have that resource. Compliance will be the main variable of the study and, in addition, the study aims to assess secondary endpoints such as quality of life (QOL).

Conclusions. NEC could increase compliance to ERAS programs, improving health outcomes and QOL perceived by the patient. The applicability in the different hospital centers could generate an opportunity to advance professionally in the nursing figure within the ERAS program. The fact of having NEC could also increase the efficiency of the program due to the cost-effectiveness of the nursing position, although this is not the object of the study. It would be applicable in improving perceived health and QOL, so it could also have an economic impact on the health system.

DETAILED DESCRIPTION:
Background. Fast-track Surgery or Enhanced Recovery After Surgery (ERAS), also called multimodal rehabilitation in Spain, constitutes the application of a series of perioperative measures and strategies aimed at those patients who undergo surgery with the objective to reduce surgical stress, promoting a better recovery of the patient by significantly reducing complications and mortality.

The ERAS programs have represented an important change in the surgical field since it opens a new line of action different from the traditional one. These protocols include a set of perioperative measures applied in a multidisciplinary way, whose advantages have been scientifically endorsed. However, these programs still face more traditional attitudes and practices, so their application is still limited today.

The Nurse ERAS Coordinator (NEC) was integrated into the multidisciplinary teams at the same time of implementation of the programs in the northern European countries, betting on their leadership and capacity from the beginning. This figure ensures that the ERAS guidelines advance in the process until their final approval and participate in the fulfillment of the protocol in the different phases. They carry out interventions based on as much evidence as possible and contribute to the collection of data for ongoing audits. In addition, they are characterized by high levels of communication skills, resourcefulness and innovation, these being key attributes of the ERAS coordinator and favoring the participation of the entire multidisciplinary team through organizational change.

Starting in the 1990s, two groups of surgeons presented different measures to improve the postoperative evolution of patients who underwent elective colorectal surgery. Both groups emphasized the importance of the information provided to the patient and its role in postoperative recovery. In Europe, specifically at the Hvidovre University Hospital in Denmark, the first group led by Kehlet emerged, who proposed different strategies to improve the postoperative period of these patients; also acting preoperatively and during surgery. Years later, the second group emerged in the United States, led by Delaney et al. from the Cleveland Clinic, who focused his studies on postoperative improvement based on the advances of the previous group, specifically in the administration of an early diet and the stimulation of early mobilization. In this way, the ERAS programs emerged.

However, it was not until 2001, when the ERAS group was formed, made up of different colorectal surgery units from 5 northern European countries (Scotland, Sweden, Denmark, Norway and the Netherlands). This group agreed on what they would call the ERAS project led by Kehlet. The recommended actions began at the moment of diagnosis and sought to recognize the individual needs of the patient to optimize their treatment before, during and after surgery.

Most of the studies whose objective has been to evaluate the efficacy of the measures that make up the ERAS program, agree that their implementation is beneficial for patients and is directly related to compliance with these measures in each of the perioperative phases.

In this sense, it is essential to consider the following key points of the program, extracted from the consensus of experts and published guides:

1. All patients participating in the protocol must start it preoperatively, which allows them a faster recovery from surgery and postoperative convalescence, minimizing physical and psychological stress.
2. The prior preparation of the patient is essential and ensures that he is in the best possible condition, identifying personal risks in the preoperative.
3. The treatment is comprehensive and includes pre, intra and postoperative measures in which the investigators act actively.
4. Patients have an active role and must take responsibility to improve their recovery.
5. Preoperative or prehabilitation period: to optimize the physical, nutritional, emotional, medical and pharmacological status of the patient; to arrive at surgery in the best possible conditions.
6. Intraoperative period: laparoscopic surgery, fluid restriction, pain control, multimodal analgesia.
7. Postoperative period: ambulation and early intake, antithrombotic measures, respiratory physiotherapy.

The implementation of ERAS programs also contributes to the improvement in the QOL perceived by the patient during the first phases of recovery. Furthermore, as a consequence, it produces a reduced general economic cost due to the decrease in the average stay in most cases.

Despite all the above, there is no evidence available that evaluates the direct impact of the NEC figure, which was implemented in 2001 in Northern Europe, the United States and Canada with a fundamental role. This is the first trial that analyzes the impact on compliance and, therefore, on health and QOL results in patients with colorectal surgery within ERAS programs.

Ethics. The study will be carried out in accordance with the Declaration of Helsinki and the Spanish laws and regulations for biomedical research. The trial protocol and patient information have been approved by the competent Ethics Committees of all participating trial centers. The data collection is part of the usual clinical practice of each participating center. For the present study, the data will be collected from the electronic medical record; therefore, the Research Ethics Committee is requested to exempt the informed consent.

During the trial, the database will not contain any identifying information about the patient. A separate document will contain the relationship of each patient with the assignment of an alphanumeric code, to which only the main researcher of the project will have access. Trials findings will be stored in accordance with Spanish data protection law (Law 15/1999 on the protection of personal data) and will be handled in strictest confidence. For protection of these data, organizational procedures are implemented to prevent distribution of data to unauthorized people.

Management of patients and Follow-up. The program was presented to the Ethics and Research Committees Clinic of both centers to, after approval, be coordinated by the NEC in BUH. NEC will be in charge of informing and training all professionals involved in any service and discipline. She will be responsible for appointing a referral from each specialty, with whom she will communicate constantly and through which all the information will be distributed through the different professionals.

Before starting the program, meetings will be convened with the heads of anesthesiology service, general and digestive surgery and nursing. The purpose of these meetings initially will be to establish synergies and align shared objectives.

Data will be collected by different professionals at each stage, but it will be the NEC who ensures and supervises the correct completion of them throughout the process. In the preadmission stage will be registered by the NEC, as well as in the immediate preoperative stage. To intraoperative level, the responsible anesthesiologist will register it. Finally, the team of surgeons will record the variables in the postoperative period. The measurement of the compliance variable will be based on the indicators of colorectal process: 17 process indicators and 2 result indicators will be evaluated following the ERAS Society audit guidelines.

Regarding the measurement of QOL, a self-administered questionnaire on the first visit of the program by the NEC, re-administering the same at 90 days postoperative: SF-12 to all patients, EORTC QLQ C30 and CR-29 in case of neoplasia.

In HGTiP, the hospital which does not have NEC, it will be the lead surgeon or head of the program who assumes this role in all the stages.

Sample size of the study. The sample size for two independent proportions (compliance), accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 103 subjects are necessary in first group and 103 in the second to find as statistically significant a proportion difference, expected to be of 0.5 in intervention group and 0.3 in control group. It has been anticipated a drop-out rate of 10%.

Statistical analysis. Descriptive methods will be used to present the distribution of variables in the study groups, with frequencies and percentages with the corresponding 95% confidence interval (CI) for categorical variables, and mean and standard deviation (SD) or median and interquartile range (25th-75th percentile) for quantitative variables. The chi-square (χ2) test will be used for the comparison of categorical variables. Clinically relevant or statistically significant variables in the bivariate analysis as well as possible confounding variables will be analyzed in a binary logistic regression model. The Mann-Whitney test will be used for the comparison of continuous variables. Also, a longitudinal analysis of variables collected at follow-up (QOL) will be performed. Statistical significance is set at P< 0.05. All analyses will be done using SPSS program, version 26.0.

Discussion. ERAS programs incorporate a series of evidence-based strategies with the aim of reducing the stress triggered by surgery and increasing functional recovery. This implies a reduction in postoperative complications, hospital stay and generates health savings. Monitoring the degree of compliance with the different strategies is necessary, not only to assess its quality and identify points for improvement, but also because the level of compliance with the program influences the patients' health results.

Despite heterogeneity in coordination and management, ERAS programs are evaluated as successful from a nurse's perspective. Continuous staff education and coordination beyond the implementation period appear to be of the utmost importance for a sustained program and the role of NEC is very important.

The available evidence suggests patients suffer no detriment to satisfaction or QOL with use of ERAS protocols, and may suffer less fatigue and return to activities sooner. The use of ERAS protocols in colorectal surgery achieves a positive influence, not only by decreasing surgical-related complications but also in terms of functional recovery, by decreasing the negative effects of surgery on patient QOL.

The main objective of this study is to demonstrate that the tertiary hospitals that integrate the NEC in the ERAS programs, obtain a higher compliance than the hospitals that do not; improving health outcomes and perceived QOL of elective colorectal surgery patients.

The investigators believe that the NEC can be a key element in the implementation of ERAS programs, commonly coordinated by surgeons and anaesthesiologists, since as described above, they are part of the implementation team and would only require a role of competencies enlarged; having more prominence in the status of projects.

In addition, the investigators consider that having this figure could lead to an improvement in the QOL perceived by the patient within the ERAS programs, due to the monitoring carried out by the ERAS Nurse Coordinator throughout the perioperative process according to the definition of its functions and the possible increase in compliance with the protocol it causes, improving health outcomes.

At the same time, lower secondary morbidity can translate into lower hospital costs (fewer stays and fewer admissions).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Candidates to elective major colorectal surgery due to benign or malignant pathology

Exclusion Criteria:

* Rejection of the patient to participate in ERAS program
* Inadequate social support that makes it difficult to comply with a discharge planned hospital
* Associated psychiatric illness, mental or organic disorders which could interfere with receiving treatments or indications about the program
* Patients with combined surgeries or simultaneous with other specialties by synchronism.
* Patients with emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Relationship between compliance to Enhanced Recovery After Surgery program and Nurse ERAS Coordinator as assessed by ERAS Society Guidelines | 30 days
  The primary endpoint is to evaluate the impact of the implementation of the Nurse ERAS Coordinator, within the ERAS program, in relation to the compliance of patients undergoing colorectal surgery in tertiary hospitals in the province of Barcelona.
  The percentage of adherence to the ERAS program will be compared in the hospital that has the Nurse ERAS Coordinator vs. the hospital that does not have that figure. The measurement will be carried out according to the process indicators proposed by the ERAS Society Guidelines.
  Wil be analyzed the relationship between protocol compliance percentage and the presence of Nurse ERAS Coordinator en each participating hospital.

SECONDARY OUTCOMES:
Quality of Life undergoing ERAS programs as assessed by SF-12 questionnaire. | 90 days
  To analyze the Quality of Life of patients undergoing ERAS program and the relationship between percentage of compliance to ERAS protocol (according to ERAS Society Guidelines) and the presence of Nurse ERAS Coordinator en each participating hospital.
  Short Form-12 (SF-12) is made up of a subset of 12 items.Each question receives a value that is later transformed into a scale from 0 to 100.Values higher or lower than 50 indicate a better or worse state of health, respectively, than the reference population.
Quality of Life undergoing ERAS programs as assessed by EORTC QLQ C30 questionnaire. | 90 days
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 is an specific questionnaire for cancer.Score between 0 and 100 is obtained.High values in the global health indicate a better quality of life,while in the symptoms scale it would indicate a decrease in quality of life.
Quality of Life undergoing ERAS programs as assessed by EORTC QLQ CR-29 questionnaire. | 90 days
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) CR-29 questionnaire includes specific questions on gastrointestinal symptoms.Minimum,maximum and scores values are the same as C30.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Jerez-Gonzalez, MSc, Principal Investigator — Hospital Universitari de Bellvitge; M.Carmen Moreno-Arroyo, PhD, Study Director — University of Barcelona; Miguel Angel Hidalgo-Blanco, PhD, Study Director — University of Barcelona
Locations (1):
- Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Kehlet H, Wilmore DW. Fast-track surgery. Br J Surg. 2005 Jan;92(1):3-4. doi: 10.1002/bjs.4841. No abstract available. PMID 15635603
- [Background] Gustafsson UO, Oppelstrup H, Thorell A, Nygren J, Ljungqvist O. Adherence to the ERAS protocol is Associated with 5-Year Survival After Colorectal Cancer Surgery: A Retrospective Cohort Study. World J Surg. 2016 Jul;40(7):1741-7. doi: 10.1007/s00268-016-3460-y. PMID 26913728
- [Background] Baimas-George M, Cochran A, Tezber K, Kirks RC, Addor V, Baker E, Martinie J, Iannitti D, Vrochides D. A 2-Year Experience With Enhanced Recovery After Surgery: Evaluation of Compliance and Outcomes in Pancreatic Surgery. J Nurs Care Qual. 2021 Apr-Jun 01;36(2):E24-E28. doi: 10.1097/NCQ.0000000000000487. PMID 32282506
- [Background] Watson DJ. Nurse coordinators and ERAS programs. Nurs Manage. 2018 Jan;49(1):42-49. doi: 10.1097/01.NUMA.0000527718.90264.89. No abstract available. PMID 29287049
- [Background] Gillissen F, Hoff C, Maessen JM, Winkens B, Teeuwen JH, von Meyenfeldt MF, Dejong CH. Structured synchronous implementation of an enhanced recovery program in elective colonic surgery in 33 hospitals in The Netherlands. World J Surg. 2013 May;37(5):1082-93. doi: 10.1007/s00268-013-1938-4. PMID 23392451
- [Background] Delaney CP, Fazio VW, Senagore AJ, Robinson B, Halverson AL, Remzi FH. 'Fast track' postoperative management protocol for patients with high co-morbidity undergoing complex abdominal and pelvic colorectal surgery. Br J Surg. 2001 Nov;88(11):1533-8. doi: 10.1046/j.0007-1323.2001.01905.x. PMID 11683754
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Anderson AD, McNaught CE, MacFie J, Tring I, Barker P, Mitchell CJ. Randomized clinical trial of multimodal optimization and standard perioperative surgical care. Br J Surg. 2003 Dec;90(12):1497-504. doi: 10.1002/bjs.4371. PMID 14648727
- [Background] Delaney CP, Zutshi M, Senagore AJ, Remzi FH, Hammel J, Fazio VW. Prospective, randomized, controlled trial between a pathway of controlled rehabilitation with early ambulation and diet and traditional postoperative care after laparotomy and intestinal resection. Dis Colon Rectum. 2003 Jul;46(7):851-9. doi: 10.1007/s10350-004-6672-4. PMID 12847356
- [Background] Gatt M, Anderson AD, Reddy BS, Hayward-Sampson P, Tring IC, MacFie J. Randomized clinical trial of multimodal optimization of surgical care in patients undergoing major colonic resection. Br J Surg. 2005 Nov;92(11):1354-62. doi: 10.1002/bjs.5187. PMID 16237744
- [Background] Khoo CK, Vickery CJ, Forsyth N, Vinall NS, Eyre-Brook IA. A prospective randomized controlled trial of multimodal perioperative management protocol in patients undergoing elective colorectal resection for cancer. Ann Surg. 2007 Jun;245(6):867-72. doi: 10.1097/01.sla.0000259219.08209.36. PMID 17522511
- [Background] Muller S, Zalunardo MP, Hubner M, Clavien PA, Demartines N; Zurich Fast Track Study Group. A fast-track program reduces complications and length of hospital stay after open colonic surgery. Gastroenterology. 2009 Mar;136(3):842-7. doi: 10.1053/j.gastro.2008.10.030. Epub 2008 Nov 1. PMID 19135997
- [Background] Serclova Z, Dytrych P, Marvan J, Nova K, Hankeova Z, Ryska O, Slegrova Z, Buresova L, Travnikova L, Antos F. Fast-track in open intestinal surgery: prospective randomized study (Clinical Trials Gov Identifier no. NCT00123456). Clin Nutr. 2009 Dec;28(6):618-24. doi: 10.1016/j.clnu.2009.05.009. Epub 2009 Jun 17. PMID 19535182
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Shanahan JL, Leissner KB. Prehabilitation for the Enhanced Recovery After Surgery Patient. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):880-882. doi: 10.1089/lap.2017.0328. Epub 2017 Jul 28. PMID 28753110
- [Background] Brooks NA, Kokorovic A, McGrath JS, Kassouf W, Collins JW, Black PC, Douglas J, Djaladat H, Daneshmand S, Catto JWF, Kamat AM, Williams SB. Critical analysis of quality of life and cost-effectiveness of enhanced recovery after surgery (ERAS) for patient's undergoing urologic oncology surgery: a systematic review. World J Urol. 2022 Jun;40(6):1325-1342. doi: 10.1007/s00345-020-03341-6. Epub 2020 Jul 9. PMID 32648071
- [Background] Watson DJ. The role of the nurse coordinator in the enhanced recovery after surgery program. Nursing. 2017 Sep;47(9):13-17. doi: 10.1097/01.NURSE.0000522018.00182.c7. No abstract available. PMID 28834927
- [Background] Balfour A, Burch J, Fecher-Jones I, Carter FJ. Understanding the benefits and implications of Enhanced Recovery After Surgery. Nurs Stand. 2019 Jul 5;34(7):70-75. doi: 10.7748/ns.2019.e11306. PMID 31468822
- [Background] Elias KM, Stone AB, McGinigle K, Tankou JI, Scott MJ, Fawcett WJ, Demartines N, Lobo DN, Ljungqvist O, Urman RD; ERAS(R) Society and ERAS(R) USA. The Reporting on ERAS Compliance, Outcomes, and Elements Research (RECOvER) Checklist: A Joint Statement by the ERAS(R) and ERAS(R) USA Societies. World J Surg. 2019 Jan;43(1):1-8. doi: 10.1007/s00268-018-4753-0. PMID 30116862
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Calderon C, Ferrando PJ, Lorenzo-Seva U, Ferreira E, Lee EM, Oporto-Alonso M, Obispo-Portero BM, Mihic-Gongora L, Rodriguez-Gonzalez A, Jimenez-Fonseca P. Psychometric properties of the Spanish version of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Qual Life Res. 2022 Jun;31(6):1859-1869. doi: 10.1007/s11136-021-03068-w. Epub 2021 Dec 20. PMID 34928470
- [Background] Arraras JI, Suarez J, Arias de la Vega F, Vera R, Asin G, Arrazubi V, Rico M, Teijeira L, Azparren J. The EORTC Quality of Life questionnaire for patients with colorectal cancer: EORTC QLQ-CR29 validation study for Spanish patients. Clin Transl Oncol. 2011 Jan;13(1):50-6. doi: 10.1007/s12094-011-0616-y. PMID 21239355
- [Background] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Background] Ban KA, Berian JR, Ko CY. Does Implementation of Enhanced Recovery after Surgery (ERAS) Protocols in Colorectal Surgery Improve Patient Outcomes? Clin Colon Rectal Surg. 2019 Mar;32(2):109-113. doi: 10.1055/s-0038-1676475. Epub 2019 Feb 28. PMID 30833859
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] ERAS Compliance Group. The Impact of Enhanced Recovery Protocol Compliance on Elective Colorectal Cancer Resection: Results From an International Registry. Ann Surg. 2015 Jun;261(6):1153-9. doi: 10.1097/SLA.0000000000001029. PMID 25671587
- [Background] Pache, B., Hübner, M., Martin, D. et al. Requirements for a successful Enhanced Recovery After Surgery (ERAS) program: a multicenter international survey among ERAS nurses. Eur Surg 53, 246-250 (2021). https://doi.org/10.1007/s10353-021-00698-9
- [Background] Leon Arellano M, Tejedor P, Guadalajara H, Ortega M, Garcia Olmo D, Pastor C. Evolution of perioperative quality of life in patients under enhanced recovery after surgery care in colorectal cancer. Rev Esp Enferm Dig. 2020 Feb;112(2):127-132. doi: 10.17235/reed.2020.6423/2019. PMID 31960699